CLINICAL TRIAL: NCT02796417
Title: Implementation of REHACOP Cognitive Training Program in Schizophrenia
Brief Title: The Efficacy of REHACOP Program in Schizophrenia
Acronym: CSrehacopSZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSMC-003-UD
Record Dates: First submitted 2016-05-13; First posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehacop group (Experimental): Cognitive rehabilitation
  Interventions: Behavioral: REHACOP
- Control group (Active Comparator): Occupational activities
  Interventions: Behavioral: Occupational activities

INTERVENTIONS:
Behavioral: REHACOP — REHACOP group consists of 90-minute-long sessions 3 days per week. Specifically, REHACOP group remediation consisted of: Attention unit (4 weeks) training sustained, selective, alternant and divided attention; Memory unit (3 weeks) focusing on visual and verbal learning, recall and recognizing memory; Language unit (3 weeks) including grammar, syntax, vocabulary, verbal fluency, verbal comprehension, abstract language; Executive functions unit (2 weeks) training cognitive planning, proverbs, analogies; and Social cognition unit (1 week) exercising theory of mind, social reasoning and moral dilemmas
  Arms: Rehacop group
Behavioral: Occupational activities — Occupational group activities conducted included drawing, gardening, reading the daily news and constructing using different materials (such as paper or wood).
  Arms: Control group

SUMMARY:
This study examined the efficacy of an integrative cognitive remediation program (REHACOP) to improve cognition, social cognition, clinical symptoms and functional outcome in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic criteria for Schizophrenia according to American Psychiatric Association's Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR)

Exclusion Criteria:

* evidence of alcohol or drug abuse in the last 30 days
* previous history of significant lack of consciousness
* mental retardation
* relevant neurological or medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in functional competence after receiving cognitive remediation | 4 months
  functional competence was measured with San Diego UCSD Performance-Based Skills Assessment- UPSA
Change in global functioning after receiving cognitive remediation | 4 months
  global functioning measured with Global Assessment of Functioning (GAF)
change in verbal memory after receiving cognitive remediation | 4 months
  Verbal memory performance was assessed with the Hopkins Verbal Learning Test-HVLT (Brandt and Benedict 2001)
change in processing speed after receiving cognitive remediation | 4 months
  Processing speed was assessed with Digit Symbol subtest from Wechsler Adult Intelligence Scale-III (Wechsler 1997)

SECONDARY OUTCOMES:
change in emotion perception after receiving cognitive remediation | 4 months
  emotion perception was assessed with Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT)
change in clinical symptoms after receiving cognitive remediation | 4 months
  Clinical symptoms was measured with Positive and Negative Syndrome Scale (PANSS)
change in social perception after receiving cognitive remediation | 4 months
  Social perception was assessed with the Social Featuring Recognition Test (SFRT)
change in theory of mind after receiving cognitive remediation | 4 months
  Theory of mind was assessed with Happe Strange Stories Test

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Ojeda, PhD, Principal Investigator — University of Deusto
Locations (1):
- University of Deusto, Bilbao, Biskai, Spain

REFERENCES:
- [Derived] Pena J, Ibarretxe-Bilbao N, Sanchez P, Uriarte JJ, Elizagarate E, Gutierrez M, Ojeda N. Mechanisms of functional improvement through cognitive rehabilitation in schizophrenia. J Psychiatr Res. 2018 Jun;101:21-27. doi: 10.1016/j.jpsychires.2018.03.002. Epub 2018 Mar 6. PMID 29525739
- [Derived] Pena J, Ibarretxe-Bilbao N, Sanchez P, Iriarte MB, Elizagarate E, Garay MA, Gutierrez M, Iribarren A, Ojeda N. Combining social cognitive treatment, cognitive remediation, and functional skills training in schizophrenia: a randomized controlled trial. NPJ Schizophr. 2016 Nov 9;2:16037. doi: 10.1038/npjschz.2016.37. eCollection 2016. PMID 27868083